CLINICAL TRIAL: NCT02795273
Title: A Combined Phase 2b/3, Randomised, Double-Blind, Placebo-Controlled, Parallel-Group, Multi-Centre Study to Assess the Efficacy and Safety of Grass-SPIRE in Subjects With Grass Pollen-Induced Allergic Rhinitis, With or Without Conjunctivitis
Brief Title: Efficacy and Safety of Grass-SPIRE Registration Study
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Decision made to stop study following availability of results from another study
Sponsor: Circassia Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TG005
Record Dates: First submitted 2016-05-05; First posted 2016-06-10 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Rhinitis; Conjunctivitis
Keywords: Rhinitis; Conjunctivitis; Grass; Allergy
MeSH Terms: conditions — Rhinitis; Conjunctivitis; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Grass-SPIRE (Experimental): Eight intradermal injections of Grass-SPIRE
  Interventions: Drug: Grass-SPIRE
- Placebo (Placebo Comparator): Eight intradermal injections of Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Grass-SPIRE
  Arms: Grass-SPIRE
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety of Grass-SPIRE compared with placebo and to evaluate the treatment effect of Grass-SPIRE on symptoms and use of rescue medication during the grass pollen season

ELIGIBILITY:
Inclusion Criteria:

* Clinical history of grass pollen-induced allergic rhinitis with or without conjunctivitis for at least 2 years
* Score of ≤ 21 on RCAT questionnaire
* Rye grass specific IgE of ≥ 0.7 kU/L
* Positive skin prick test to Rye grass whole allergen extract

Exclusion Criteria:

* History or findings of significant disease
* Asthma requiring GINA Step 3 or higher treatment
* History of severe drug allergy, severe angioedema or systemic allergic reaction
* Course of short-duration allergy-specific immunotherapy or more than 3 months treatment with long-duration allergen immunotherapy within 5 years
* Contraindications for administration of epinephrine

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Combined Score of symptoms and allergy medication | Approximately 66 weeks
  Measurement of subject allergy symptoms (eg sneezing, watery eyes) and use of allergy medication
Safety of Grass-SPIRE | Approximately 66 weeks
  Measurement of adverse events

SECONDARY OUTCOMES:
Symptom Scores | Approximately 66 weeks
  Categorical scores of allergy symptoms (eg sneezing, watery eyes) as assessed by subjects
Rescue Medication Use | Approximately 66 weeks
  Use of allergy medication to help allergy symptoms
Quality of Life | Approximately 66 weeks
  Assessment of Quality of Life measured by responses to a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: David Bernstein, MD, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - Canton, Ohio
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Undecided